CLINICAL TRIAL: NCT01163175
Title: Study of the Impact of Trans Fatty Acids From Dairy Products n Cardiovascular Risk Factors
Brief Title: Study of the Impact of Trans Fatty Acids From Dairy Products on Cardiovascular Risk Factors
Acronym: TRANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Dairy Farmers of Canada (Other); Novalait Inc (Unknown)
Responsible Party: Benoît Lamarche, PhD, Institute of Nutraceutical and Functional Foods (INAF), Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INAF-2005-233
Record Dates: First submitted 2010-07-09; First posted 2010-07-15 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2010-07

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular disease; Trans fatty acids; Ruminant; Blood lipids
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Ruminant trans fats — Consumption of the 4 experimental diets:
  1. a diet rich in ruminant TFA (8 g/day);
  2. a diet moderately rich in ruminant TFA (4 g/day);
  3. a diet rich in industrial TFA (8 g/d);
  4. a control diet (minimal dietary TFA of industrial and ruminant sources).

SUMMARY:
The majority of trans fatty acids consumed by the general population is derived from products that have been formulated using significant amount of hydrogenated vegetable oil (the so-called industrial trans fat). Fat from ruminants also contains small amounts of trans fatty acid, which contribute, although to a smaller extent, to the total dietary intake of trans fatty acids in the general population. The negative impact of consuming industrial trans fat on health, particularly on cardiovascular disease, is being increasingly recognized. Based on data available to date, it is currently not possible to conclude if effects of ruminants and industrial trans fatty acid on cardiovascular risk are different. There is therefore an urgent need for a study that compares the impact of naturally occurring trans fatty acids such as those from dairy products and of trans fatty acids form industrial sources on cardiovascular risk factors as well as their mechanisms of action.

The general objective of the study is to investigate the impact of naturally occurring trans fatty acids from dairy products (mainly vaccenic acid) on plasma cholesterol levels and other risk factors for cardiovascular disease.

DETAILED DESCRIPTION:
The proposed research will be undertaken as a double-blind randomized cross-over study according to a Latin Square design, with participants being subjected to 4 consecutive isocaloric diets in random order lasting 4 weeks each. No stratification is considered since the population recruited will be relatively homogeneous. The 4 experimental diets are: 1- a diet rich in ruminant TFA (8 g/day); 2- a diet moderately rich in ruminant TFA (4 g/day); 3- a diet rich in industrial TFA (8 g/d); 4- a control diet (minimal dietary TFA of industrial and ruminant sources). The source of ruminant TFA will come from butter and cream obtained after having modified the regimen of lactating cows in a fashion similar to the one used to increase the levels of conjugated linoleic acid (CLA) in milk fat. Hydrogenated margarine will be used as the main source of industrial TFA. Finally, a butter obtained from cows producing the lowest levels of ruminant fat will be used to formulate the control diet (minimal dietary TFA). All diets will be identical in terms of menus, calories and macronutrient composition with the exception of TFA sources and levels. Minor differences in the levels of total saturated, monounsaturated and polyunsaturated fatty acids will be matched across diets by adding various vegetable and animal oils. The macronutrient composition of each meal and thus of the entire day is very similar across all 4 diets. Based on a 2500 kcal/day regimen, an intake of TFA of 8 g/d and 4 g/d will represent 72 kcal/day and 36 kcal/day respectively (3% and 1.5% of energy intake). The 4 experimental diets will be formulated so that the percentage of daily calories from fat (36%), carbohydrates (50%) and proteins (14%) will meet most of the dietary recommendations of the American Heart Association and the NCEP for primary prevention of CVD, with the exception of SAT (slight excess) and fibers (slight deficit). The slight excess in SAT fat cannot be avoided since we are using butter as the primary source of ruminant TFA. The cholesterol content of the experimental diet will not exceed 300 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* LDL-Cholesterol concentration <3.4 mmol/L
* Stable body weight (+/- 2 kg) for 6 months before the beginning of the study
* Smoking or not

Exclusion Criteria:

* Previous history of cardiovascular disease, type 2 diabetes and monogenic dyslipidemia
* Subjects taking medications for hyperlipidemia or hypertension
* Endocrine disorders
* Body mass index > 30 kg/m2
* Food allergies
* Men with extreme nutritional habits such as vegetarism or alcohol consumption > 2 drinks/day
* Elite athletes

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2006-05; Primary Completion 2007-07 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Plasma LDL-Cholesterol concentrations | At the beginning and the end of the 4 for-week diets

SECONDARY OUTCOMES:
Blood lipids and apolipoproteins levels (Total cholesterol, HDL-Cholesterol, Triglycerides, Apo A1, Apo B) | At the beginning and the end of the 4 for-week diets
Markers of inflammation (C-reactive protein) | At the beginning and the end of the 4 for-week diets
Blood pressure | At the beginning and the end of the 4 for-week diets
Anthropometric measures (waist and hip circumferences) | At the beginning and the end of the 4 for-week diets
Surrogates of cholesterol absorption and synthesis | At the beginning and the end of the 4 for-week diet

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Lamarche, PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutraceutical and Functional Foods (INAF), Laval University, Québec, Quebec, Canada